CLINICAL TRIAL: NCT05905900
Title: Emergent Intravenous Dye Preparation for Acute Stroke Patients With a History of Intravenous Dye Allergy
Brief Title: Emergent Prep for IV Dye in Acute Stroke Patients With Allergy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Global Neurosciences Institute (Other)
Collaborators: Drexel University College of Medicine (Other)
Responsible Party: Principal Investigator, Erol Veznedaroglu, President and CEO Global Neurosciences Institute, Global Neurosciences Institute
Other Study IDs: IVDyeAllergy
Record Dates: First submitted 2023-06-07; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Stroke; Dye Allergy
Keywords: Stroke; Emergent IV Dye Prep; Dye Allergy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Emergent IV Dye Preparation & Administration: The emergent IV dye drug trio is administered and followed immediately by Computed Tomography (CT) Angiography and/or CT Perfusion.
  Interventions: Combination Product: Emergent IV Dye Preparation

INTERVENTIONS:
Combination Product: Emergent IV Dye Preparation — Diphenhydramine 50 mg IV once, famotidine 20 mg IV once, and dexamethasone 10 mg IV once

SUMMARY:
Our institution implemented a protocol to administer an emergent IV dye preparation for stroke alert patients requiring advanced neuroimaging. The emergent IV dye preparation consists of diphenhydramine 50 mg IV once, famotidine 20 mg IV once, and dexamethasone 10 mg IV once, followed immediately by Computed Tomography (CT) Angiography and/or CT Perfusion.

DETAILED DESCRIPTION:
Patients with documented IV dye allergy were given emergent dye preparation immediately prior to advanced neuroimaging that consisted of three drugs: diphenydramine 50 mg IV, famotidine 20 mg IV, and dexamethasone 10 mg IV. In contrast, elective dye preparation commonly done in non-emergent or outpatient settings is separated into two different options. The first option is for a patient to take Prednisone 50 mg three times prior to the study: one tablet by mouth 13 hours prior, one tablet by mouth seven hours prior, and the last tablet by mouth one hour prior to the study. The second option is for the patient to be prescribed dexamethasone 4 mg or 6 mg dispensed four times: two tablets by mouth 12 hours prior to the study and 2 tablets by mouth one hour prior to the study. If the patient is prescribed dexamethasone, they also take famotidine 150 mg and diphenhydramine 50 mg, both drugs by mouth 12 hours prior and one hour prior to the study.

To evaluate the relationship between dye allergy and any adverse reactions, our study's inclusion criteria consisted of all stroke alert patients from 2021-2022 who required advanced neuroimaging of CTP/CTA and received emergent IV dye preparation. Exclusion criteria included patients who reported dye allergies specific to airway edema or anaphylaxis. A retrospective chart review was done to evaluate stroke patient's stated allergies, the number of patients that received emergent IV dye preparation, and any adverse reactions despite the emergent IV dye preparation. Data was then analyzed to determine if there was a relationship between prior contrast dye allergy and allergic reactions that occurred after emergent IV dye administration.

ELIGIBILITY:
Inclusion Criteria: Stroke alert patients that required advanced neuroimaging of CTP/CTA and received emergent IV dye preparation -

Exclusion Criteria: patients who reported dye allergies specific to airway edema or anaphylaxis

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Stroke alert patients with a history of dye allergies.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Adverse Reactions | 24 Hours
  Unwanted side effects of medication administration, including but not limited to itching, rash, mild shortness of breath etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Philadelphia, Pennsylvania, United States